CLINICAL TRIAL: NCT02167009
Title: Phase II, Single Arm Prospective Study to Evaluate Safety and Efficacy of Prostate Artery Embolization in Patients With Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia and Prostate Size Greater Than 90 Grams
Brief Title: Benign Prostatic Hyperplasia and Prostate Size Greater Than 90 Grams
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGH0003
Record Dates: First submitted 2014-05-07; First posted 2014-06-18 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: ARTERY EMBOLIZATION; BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate Artery Embolization (Experimental): Embospheres microspheres
  Interventions: Device: Embosphere Microspheres

INTERVENTIONS:
Device: Embosphere Microspheres — Embosphere Microspheres are indicated for use in embolization of arteriovenous malformations, hypervascular tumors, and symptomatic uterine fibroids.

SUMMARY:
Study to evaluate Prostate Artery Embolization for the treatment of lower urinary track symptoms due to Benign Prostatic Hyperplasia and Prostate Size Greater Than 90 Grams.

DETAILED DESCRIPTION:
This is a phase II, single center, prospective, single arm, investigational study to evaluate the safety and efficacy of prostate artery embolization (PAE) for treatment of severe lower urinary tract symptoms (LUTS) related to BPH in patients with prostate size greater than 90 grams that either refuse surgical treatment or are considered poor candidates for traditional surgical therapy.

30 patients will be enrolled in the single treatment arm with follow-up for no less than 12 months.

The study will involve a screening period in which patient eligibility will be determined. Once eligibility is confirmed, patients will receive PAE with Embosphere Microspheres within 4 weeks of screening and transrectal ultrasound. After treatment, patients will return for follow-up visits at 1 month, 3 months, 6 months, and 12 months post PAE. At each of these visits, patients will complete IPSS and IIEF questionnaires, undergo a physical exam, and perform a medication review. Repeat TRUS and urodynamic testing will be performed at the 6 month and 12 month post PAE follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 50-85 years
* Patient has signed informed consent
* Patient has experienced lower urinary tract symptoms (LUTS) for at least 1 year prior to study enrollment
* Patient has a prostate size larger than 90g as measured by transrectal ultrasound (TRUS)
* Patient has an IPSS score greater than or equal to 13
* Patient has a peak urine flow rate < 12 mL/sec
* Patient either:
* Refuses surgical treatment
* Is considered high risk for surgical treatment
* Patient is either:
* Refractory to medical treatment
* Contraindicated for medical treatment
* Patient must meet ONE of the following criteria:
* Baseline PSA ≤ 2.5ng/mL
* Baseline PSA > 2.5 ng/mL and ≤ 10 ng/mL AND free PSA ≥ 25% of total PSA (no biopsy required)
* Baseline PSA > 2.5 ng/mL and ≤ 10 ng/mL AND free PSA < 25% of total PSA AND negative prostate biopsy result (minimum of 12 core biopsy) within 12 months
* Baseline PSA >10 ng/mL AND negative prostate biopsy result (minimum of 12 core biopsy) within 12 months

Exclusion Criteria:

* History of prostate or bladder cancer, or currently being evaluated for cancer
* History of prostate or bladder cancer, or currently being evaluated for cancer
* Patient has taken alpha blockers within 4 weeks of screening
* Patient has experienced an irregular voiding pattern despite medical management with a stable 5-alpha reductase inhibitor dosage for 3 months or longer
* History of open prostate surgery, radiofrequency, or microwave therapy
* Previous open bladder or rectosigmoid colon surgery
* TURP within the last two years
* Patient has nodularity or induration detected upon digital rectal examination (DRE)
* Neurogenic bladder or other neurological disorder impacting bladder function
* Urethral stricture, bladder neck contracture, other potentially confounding bladder pathology, bladder disease, or confounding urethral pathology
* Acute urinary retention requiring an indwelling catheter
* Bladder atonia
* Active prostatitis or urinary tract infection
* Cystolithiasis within the past 3 months
* Serum creatinine >1.7mg/dL
* Coagulation disturbances not normalized by medical treatment
* Iodinated contrast allergy not controlled with 24-hour steroid preparation
* History of gelatin allergy
* History of pelvic irradiation
* History of severe peripheral vascular disease or known major iliac arterial occlusive disease
* History of smoking greater than 30 pack-years
* Interest in future fertility
* Significant cardiac or respiratory disease that the Investigator believes puts the patient at risk for a complication during the procedure
* Any other risks or factors that the Investigator believes puts the patient at risk for a complication during the procedure

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of BPH symptoms as assessed by the IPSS at 12 months post PAE. | Safety will be evaluated throughout the initial 12 months of the study by assessing adverse events and findings on physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Davis, MD, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States